CLINICAL TRIAL: NCT01292343
Title: Effect of a Triclosan Containing Dentifrice on Oral Bacteria and Postoperative Complications Following Third Molar Surgery
Brief Title: Triclosan Toothpaste and Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Yanfang Ren, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UREDC3rd
Record Dates: First submitted 2011-02-04; First posted 2011-02-09 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Dry Socket; Wound Infection
Keywords: third molars; triclosan; toothpaste; dry socket; wound infection
MeSH Terms: conditions — Dry Socket; Wound Infection | interventions — hydrated silica gel-based toothpaste; Triclosan; Dentifrices; Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Colgate Total Toothpaste — Toothbrushing with Colgate Total Toothpaste
  Other Names: triclosan; dentifrice
Other: Colgate Regular Toothpaste — Toothbrushing with Colgate regular toothpaste
  Other Names: fluoride; dentifrice

SUMMARY:
Triclosan containing dentifrices are effective in the prevention of inflammatory complications following third molar surgery through reducing preoperative oral bacteria load.

DETAILED DESCRIPTION:
This study may provide evidence on the effect of triclosan containing dentifrice on oral bacteria and oral inflammation prior to third molar surgery, and on the incidence of inflammatory complications after the surgery. If proven effective, dentifrice containing triclosan may be recommended prior to tooth extractions and replace antibiotics and other antimicrobial products as a prophylactic procedure before oral surgery procedures.

ELIGIBILITY:
Inclusion Criteria:

* must include at least one mandibular third molar with partial or full bony impaction
* no sign of active pericoronal (around the crown) infections
* must have not taken antibiotics for any reason in the past 30 days
* must be healthy and between 18 and 35 years of age
* must be able to read and sign an informed consent

Exclusion Criteria:

* Subjects with systemic diseases and pregnant or lactating women
* Subjects with advanced periodontal diseases or having two or more untreated caries lesions
* Subjects who cannot read and sign an informed consent
* Subjects with signs of pericoronal infections

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
dry socket | 3 to 7 days
  Development of dry socket (alveolar osteitis) 3 to 7 days after tooth extraction

SECONDARY OUTCOMES:
wound infection | 3 to 7 days
  Development of tooth extraction wound infection 3 to 7 days after extraction

CONTACTS AND LOCATIONS:
Overall Officials: Yanfang Ren, DDS, MPH, Principal Investigator — University of Rochester Eastman Dental Center
Locations (1):
- University of Rochester Eastman Dental Center, Rochester, New York, United States